CLINICAL TRIAL: NCT01424774
Title: A Prospective Study to Estimate Inadvertent Radiation Exposure From Strontium Isotopes in Patients Who Have Undergone CardioGen-82® PET MPI Scanning
Brief Title: Prospective Evaluation of Strontium in Patients After CardioGen-82 PET MPI Scanning
Status: Completed | Type: Observational
Sponsor: Bracco Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: CGEN-105
Record Dates: First submitted 2011-08-25; First posted 2011-08-29 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-08

CONDITIONS: Radiation Exposure
Keywords: Radiation Exposure; Rubidium 82; Strontium 82; Strontium 85

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: CardioGen-82 — CardioGen-82 is not administered to patients in this study, however to be able to qualify for enrollment, the patients must have received CardioGen previously

SUMMARY:
This study will be performed at clinical sites that have administered CardioGen-82® to patients from January to July 2011. The patients enrolled(i.e., "target date patients") will be all those who were dosed at the end of use of the CardioGen-82® generators on the last day of generator use from the generator that was used immediately prior to the recalled generator (i.e., "target date generators"). These are not patients who received drug eluted from the recalled generator. Of these patients, it is planned that 100 patients will be entered in this trial.

DETAILED DESCRIPTION:
This clinical study protocol will use a three tier approach consisting of the following examinations:

1. Patient examination with Survey Meter: Patients who agree to be tested at the clinical sites will be first evaluated using a survey meter. In those patients in whom radiation count is ≥ 2 times above background count using a standard survey meter, the presence of Sr-82 and/or Sr-85 will be assessed through a quantitative reading from a calibrated portable isotope identifier.
2. Patient examination with Portable Isotope Identifier: This examination will be done by use of a portable isotope identifier, which will be supplied by the Sponsor to the study sites. An assessor, independent to the study site, will perform the examination. In those patients whose radiation count is ≥ 2 times above background count using a standard survey meter, the presence of Sr-82 and/or Sr-85 will be assessed through a quantitative reading from a calibrated portable isotope identifier. The reading will be forwarded along with the date of the reading, the date of the patient's CardioGen-82® scan, and the total dose of CardioGen-82® administered to the patient, to an independent medical expert, independent to the study site, who will back-calculate an estimated dose of Sr-82 and/or Sr-85 from these data.
3. Patient examination at Oak Ridge National Laboratory: Any patient whose estimated dose of Sr-82 exceeds the specified limit of 0.02 microcuries per mCi Rb-82 administered, and/or whose estimated dose of Sr-85 exceeds the specified limit of 0.2 microcuries per mCi Rb-82 administered, will be asked to travel to Oak Ridge National Laboratory in Tennessee, for accurate whole body scanning. Scan data from Oak Ridge National Laboratories will be analyzed by one or more independent medical experts to accurately back-calculate exposure to Sr-82 and/or Sr-85, and to estimate health hazard for the patient.

ELIGIBILITY:
Inclusion Criteria:

Enroll a patient in this study if the patient meets the following inclusion criteria:

* Male or female
* Gave informed consent to participate in the study
* Received CardioGen-82® that had been eluted from the generator on the last usage day the generator was used prior to the generator that was recalled.

Exclusion Criteria:

* Exclude a patient from this study if the patient has previously been enrolled in and completed this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population would come from sites who administered CardioGen-82® during the time period of January 2011 to July 2011. The patient population is expected to be patients (i.e., target date patients) who were administered Caridogen-82 that had been eluted from the generator on the last usage day the generator was used prior to the generator that was recalled (i.e., target date generator). It is planned to enroll 100 patients in this study. Each site that agrees to participate will be encouraged to enroll at least 1 patient. Depending on the number of sites agreeing to participate, the enrollment time frame may be extended to include the last 3 to 5 days of generator usage.
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2011-09; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Determination of radiation exposure from Sr-82/Sr-85 | on average within 24 hours
  To determine radiation exposure from Sr-82 and/or Sr-85 in "target date patients" administered CardioGen-82® for PET MPI. "Target date patients" are defined as patients who were administered CardioGen-82® eluted on the last day of generator use from the generator that was used immediately prior to the recalled generator (i.e., "target date generator").
Determination of extent of Sr-82/Sr-85 exposure, if positive exposure is detected | within 2 weeks
  To determine the extent of the Sr-82/Sr-85 exposure, in the subset of patients with positive testing exceeding the specified threshold for the breakthrough of Sr-82/Sr-85, by performing whole body scanning at Oak Ridge National Laboratory for eventual health hazard assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Sireci, M.D., Study Director — Bracco Diagnostics, Inc
Locations (1):
- Bracco Diagnostics, Inc., Princeton, New Jersey, United States